CLINICAL TRIAL: NCT05633940
Title: The Effects of Primary Care Behavioral Health in Primary Care in Sweden
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Collaborators: Region Jönköping County (Other Government); Region Örebro County (Other)
Responsible Party: Principal Investigator, Hanna Israelsson Larsen, Adjunct Senior Lecturer/resident physician in general medicin, Region Östergötland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-05572
Record Dates: First submitted 2021-04-21; First posted 2022-12-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Primary Health Care; Mental Disorder; Behavioral Symptoms
MeSH Terms: conditions — Mental Disorders; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation (Experimental): The centers that implement PCBH.
  Interventions: Behavioral: Implementation of the service delivery model primary care behavioral health
- No implementation (No Intervention): Control centers that do not implement PCBH.

INTERVENTIONS:
Behavioral: Implementation of the service delivery model primary care behavioral health — The research project will study a real-world implementation of PCBH in routine primary care. The implementation is facilitated by a regional implementation group of psychologists with special training in PCBH. The active implementation period for each intervention center is 12 months, where continuous support, materials and training are offered by the implementation group.
  Arms: Implementation

SUMMARY:
The novel multi-professional service delivery model "Primary Care Behavioural Health" (PCBH) has been suggested as an effective way to integrate behavioural health services into routine primary care to overcome the growing problems with psychosocial and mental health problems in primary care. In this multicenter mixed-methods pragmatic clinical trial, the implementation of PCBH in routine primary health care in a region in Sweden is investigated.

DETAILED DESCRIPTION:
Psychosocial and mental health problems is a growing public health concern and challenge for primary care where resources are scarce. The multi-professional novel service delivery model "Primary Care Behavioural Health" (PCBH) has been suggested as an effective way to integrate behavioural health services into routine primary care. The model offer high accessibility to brief interventions, is clinically intuitively attractive and has been disseminated in primary care organizations globally, as well as in Sweden. However, more research is needed on its effect and implementation in routine care. The objective is to investigate the effect of the new service delivery model PCBH on organization- staff- and patient outcomes, and to investigate the implementation of PCBH in terms of how and to which degree the new way of working is normalised in practice routines. This multicenter mixed-methods interventional study is designed as a controlled pragmatic clinical trial. The effect of PCBH will be investigated on organizational, staff and patient levels. Variables include waiting lists, symptoms, medication prescriptions, quality of life and working environment aspects. Study participants will be patients, staff and managers at the included primary care centers. Implementation of PCBH will be investigated regarding the implementation process and degree of implementation. Data will be both qualitative (individual interviews) and quantitative (registers, biomarkers and questionnaires). At least 24 intervention centers will be compared to an equal number of control centers. The research project will be conducted in several regions in Sweden during a period of 4 years. PCBH seems to offer a solution the challenges in modern primary care, but evidence is low. This study will provide much-needed clinically meaningful data regarding PCBH that hopefully could be used for future development of primary healthcare.

ELIGIBILITY:
Patients:

Inclusion Criteria, one of following:

* Adult patients who seek care for mental health problems at a participating centre,
* Adult patients who have received any following International Classification of Diseases diagnose: F00-F99, Z56, Z73
* Adult patients who are prescribed any psychotropic drugs with ATC codes: N05A-C, N06A) at a participating centre.
* Adult patients who has an appointment to a behavioral health consultant at a participating centre.

Exclusion Criteria:

• Not capable to leave informed consent.

Medical staff:

Inclusion Criteria:

• Health care professionals employed at a participating centre.

Exclusion Criteria:

• Temporarily hired personnel, e.g. hired doctors or nurses on weekly basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accessibility at the health care center, measured in number of visits | Baseline to 24 months.
  Number of visits to health care professionals treating patients for mental health issues (i.e. behavioral health consultants and physicians).
Functional level of the patients. | Baseline to 24 months.
  Measured by Sheehan disability scale.
Work environment among the medical staff | Baseline to 24 months.
  Measured by the COPSOQ III questionnaire , which is an instrument that measures psychosocial factors, stress, and the well-being of employees.
Experience of primary care behavioral health among the medical staff | Baseline to 24 months.
  Data will be collected through qualitative interviews.

SECONDARY OUTCOMES:
Accessibility at the health care center, measured in waiting times. | In total 3 years: one year before baseline (baseline: when implementation starts), thereafter during 2 year from baseline.
  Waiting times to first visit to health care professionals treating patients for mental health issues (i.e. behavioral health consultants and physicians).
Quality of life of the patients. | 2 years from baseline (first visit to a health care professional due to a mental health issue, therafter after 6, 12 and 24 months).
  Measured by Euroqol 5 dimensions 5 levels, on a scale from 1 to 5 on each item where 1 means no problems and 5 means severe problems.
Symptoms of anxiety in the patients. | 2 years from baseline (first visit to a health care professional due to a mental health issue, therafter after 6, 12 and 24 months).
  Measured by Generalised Anxiety Disorder Assessment (GAD-7), on a scale from 0-21, where higher points means higher risk for anxiety.
Symptoms of depression in the patients | 2 years from baseline (first visit to a health care professional due to a mental health issue, therafter after 6, 12 and 24 months).
  Measured by the patient health questionnaire (PHQ-9) on a scale from 0-27, where higher points means higher risk for depression.
Referrals to psychiatric care | In total 3 years: one year before baseline (baseline: when implementation starts), thereafter during 2 year from baseline.
  The number of patients with mental health issues who are referred to psychiatric specialist care.
Work commitment among the medical staff | 2 years in total: at baseline, therafter at 6, 12 and 24 months.
  Measured by the Utrecht Work Engagement Scale, where higher points mean higher work engagement.
Exhaustion among the medical staff | 2 years in total: at baseline, therafter at 6, 12 and 24 months.
  Measured by the Karolinska exhaustion disorder scale (KEDS), where higher points indicate higher risk for exhaustion disorder.
Fidelity to the core components among the medical staff | 2 years in total: at baseline, therafter at 6, 12 and 24 months.
  Measured by a questionnaire incorporating typical features of work according to primary care behavioral health.
Medical treatment of patients due to mental health issues | In total 3 years: one year before baseline (baseline: when implementation starts), thereafter during 2 year from baseline.
  Number of patients who are prescribed psychotropic drugs (ATC codes: N05A, N05B, N05C and N06A).
Sick leave of patients due to mental health issues | In total 3 years: one year before baseline (baseline: when implementation starts), thereafter during 2 year from baseline.
  Number of patients who are on sick leave due to mental health issues (defined as sick leave due to one or more F- or Z-diagnoses according to the International Classification of Diseases (ICD-10) codes in the F00-F99, Z56, Z63 and Z73 sections.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna I Larsen, PhD, Principal Investigator — region östergötland/Primärvårdscentrum/Vårdcentralen Cityhälsan centrum
Locations (1):
- Primärvårdscentrum, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared with other researchers.

REFERENCES:
- [Derived] Larsen HI, Thomas K, Nordgren LB, Ruiz ES, Koshnaw K, Nilsen P. Implementing primary care behavioral health in Swedish primary care - study protocol for a pragmatic stepped wedge cluster trial. BMC Prim Care. 2024 Aug 20;25(1):310. doi: 10.1186/s12875-024-02515-0. PMID 39164634